CLINICAL TRIAL: NCT01116193
Title: A Phase II, Multi-center, Open-label, Repeat-dose Study of Lenalidomide (Revlimid ®) Plus Low-dose Dexamethasone in Patients With Refractory B Cell Lineage Acute Lymphoblastic Leukemia or in Relapse After 2 Lines of Treatment
Brief Title: Repeat-dose Study of Lenalidomide (Revlimid ®) Plus Dexamethasone in Patients With Lymphoblastic Leukemia
Acronym: RV-405 LAL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut de Cancérologie de la Loire (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-01b; 2009-009372-13 (EudraCT Number)
Record Dates: First submitted 2010-04-26; First posted 2010-05-04 (Estimated); Last update posted 2017-09-14 (Actual); Status verified 2011-01

CONDITIONS: Leukemia, Lymphoid; Precursor B-Cell Lymphoblastic Leukemia-Lymphoma
Keywords: antileukemic therapy; lymphoblastic leukemia; lenalidomide; dexamethasone
MeSH Terms: conditions — Leukemia, Lymphoid; Precursor B-Cell Lymphoblastic Leukemia-Lymphoma; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Lenalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Lenalidomide plus dexamethasone — Lenalidomide 25 mg p.o. once daily on days 1-21 plus Dexamethasone 40 mg p.o. once daily on days 1, 8, 15, and 22 of each 28-day cycle (4-weeks cycles) until CR achievement, progression of disease or intolerable toxicity
  Other Names: Revlimid ®, 25mg

SUMMARY:
The study objectives are to evaluate the safety and efficacy of the oral administration of lenalidomide in combination with dexamethasone in the treatment of adult patients with refractory or relapsed non-Ph+ B-cell lineage acute lymphoblastic leukemia (ALL).

DETAILED DESCRIPTION:
The study consists of two periods, an initial treatment period and an extended treatment period. Patients who meet all eligibility criteria will receive: Lenalidomide 25 mg p.o. once daily on days 1-21 plus Dexamethasone 40 mg p.o. once daily on days 1, 8, 15, and 22 of each 28-day cycle (4-weeks cycles) until CR achievement, progression of disease or intolerable toxicity. The daily dose of Lenalidomide and that of Dexamethasone will remain fixed. No dose adaptations are allowed according to the hematologic toxicity. However, in case of non-hematologic grade > 2 toxicity, the next cycle may be delayed up to 21 days after the onset of the event until the adverse event has returned to baseline or ≤ grade 1. Patients may be allowed to receive a pre-treatment with high doses of dexamethasone for initial hyperleukocytosis at the discretion of the investigator. The use of hematopoietic growth factor (HGF) during the initial or extended treatment period is also let at the discretion of the investigator. At the end of the initial treatment period, all responding patients (without HLA compatible donor) or patients showing sufficient clinical activity will be allowed to receive extended treatment with cycles identical to the first cycle. Patients may continue to receive treatment as long as the patient is tolerating the treatment well and the patient's physician believes the patient is receiving some benefit. The severity of adverse events will be graded according to the World Health Organization (WHO) criteria. Any life-threatening adverse effects that are observed during the initial or extended treatment period, which are possibly or probably related to study drug, will require the subject to discontinue study treatment.

ELIGIBILITY:
Inclusion Criteria:

* Documented B-cell lineage acute lymphoblastic leukemia (non-Philadelphia positive chromosome), which under WHO guidelines is now referred to as precursor B-lymphoblastic leukemia/lymphoma.
* Must have failed to at least two treatment regimens for B lineage ALL or must be refractory to chemotherapy. The inclusion of a patient with Ph+ ALL can be possible after contacting the principal investigator in presence of a T315I mutation and absence of investigational trial targeting this abnormality.
* Performance status of ≤ 2 by Eastern Cooperative Oncology Group (ECOG) criteria.
* Any age ≥ 18 years is allowed.
* Life expectancy of at least 3 months.
* Adequate liver function (aspartate transaminase [AST] and/or alanine transaminase [ALT] not > 3 times upper limits of normal).
* Adequate kidney function (calculated creatinine clearance > 50 ml/min).
* Signed informed consent prior to start of any study-specific procedures.
* The patients refusing the preservation of their biological samples can however participate in the study.
* All subjects must

  * Agree to abstain from donating blood while taking study drug therapy and for one week following discontinuation of study drug therapy.
  * Agree not to share study medication with another person and to return all unused study drug to the investigator

Female subjects of childbearing potential must :

* Understand that the study medication is expected to have a teratogenic risk
* Agree to use, and be able to comply with, effective contraception without interruption, 4 weeks before starting study drug, throughout the entire duration of study drug therapy (including dose interruptions) and for 4 weeks after the end of study drug therapy, even if she has amenorrhoea. This applies unless the subject commits to absolute and continued abstinence confirmed on a monthly basis. The following are effective methods of contraception

  * Implant
  * Levonorgestrel-releasing intrauterine system (IUS)
  * Medroxyprogesterone acetate depot
  * Tubal sterilization
  * Sexual intercourse with a vasectomised male partner only; vasectomy must be confirmed by two negative semen analyses
  * Ovulation inhibitory progesterone-only pills (i.e., desogestrel)
  * If not established on effective contraception, the female subject must be referred to an appropriately trained health care professional for contraceptive advice in order that contraception can be initiated
* Understand that even if she has amenorrhea, she must follow all the advice on effective contraception.
* Understand the potential consequences of pregnancy and the need to rapidly consult if there is a risk of pregnancy
* Agree to have a medically supervised pregnancy test with a minimum sensitivity of 25 mIU/mL on the day of the study visit or in the 3 days prior to the study visit once the subject has been on effective contraception for at least 4 weeks. This requirement also applies to women of childbearing potential who practice complete and continued abstinence. The test should ensure the subject is not pregnant when she starts treatment
* Agree to have a medically supervised pregnancy test every 4 weeks including 4 weeks after the end of study treatment, except in the case of confirmed tubal sterilization.

Criteria for women of non-childbearing potential

A female subject or a female partner of a male subject is considered to have childbearing potential unless she meets at least one of the following criteria:

* Age ≥ 50 years and naturally amenorrhoeic for ≥ 1 year (Amenorrhoea following cancer therapy does not rule out childbearing potential.)
* Premature ovarian failure confirmed by a specialist gynaecologist
* Previous bilateral salpingo-oophorectomy, or hysterectomy
* XY genotype, Turner syndrome, uterine agenesis.

Male subjects must

* Agree to use condoms throughout study drug therapy, during any dose interruption and for one week after cessation of study therapy if their partner is of childbearing potential and has no contraception.
* Agree not to donate semen during study drug therapy and for one week after end of study drug therapy.

Exclusion Criteria:

* Active serious infection not controlled by oral or intravenous antibiotics.
* Treatment with any investigational antileukemic agent or chemotherapy agent in at least 7 days prior to study entry and lack of full recovery from side effects due to prior therapy independent of when that therapy was given.
* Rapidly progressive disease with compromised organ function judged to be life-threatening by the Investigator.
* Patients with clinical evidence of active central nervous system (CNS) disease.
* Pregnant and/or lactating female.
* Patients with known human immunodeficiency virus (HIV) infection.
* Patients with known active hepatitis B and/or hepatitis C infection.
* Hypersensitive or intolerant to any component of the study drug formulation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-01; Primary Completion 2012-07 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Disease-Free survival (DFS) | 2 years

SECONDARY OUTCOMES:
Time to response | 28 days
Duration of response | 2 years
To determine quality of life (QOL): European Organization for Research and Treatment of Cancer QOL questionnaire for patients with cancer (EORTC QLQ-C30) | All 28 days
Progression-free survival | 2 years
Feasibility of stem cell transplantation (SCT), in case of response, after one or more cycles of lenalidomide plus dexamethasone therapy | all 28 days
Safety of lenalidomide plus dexamethasone: adverse events (type, frequency, severity of adverse events, and relationship of adverse events to study drug). | All 28 days
To assess the efficacy of lenalidomide plus low-dose dexamethasone: complete response (CR), complete response without platelets (CRp), partial response (PR), and overall response (CR + CRp + PR). | 1, 8, 15, and 22 of each 28-day cycle (4-weeks cycles) and after treatment, patients will be seen at least twice weekly until they attain a CR
Overall survival | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuelle Tavernier, MD, Principal Investigator — Institut de Cancérologie de la Loire
Locations (4):
- France (4):
  - CHU de Clermont-Ferrand, Clermont-Ferrand
  - Hôpital Michallon, Grenoble
  - Hôpital Edouard Herriot, Lyon
  - Institut de Cancerologie de la Loire, Saint-Priest-en-Jarez